CLINICAL TRIAL: NCT05599217
Title: Association Between Dietary Factors and Chronic Subdural Hematoma: a Multicenter Case-control Study
Brief Title: Association Between Dietary Factors and Chronic Subdural Hematoma (DISH)
Acronym: DISH
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Weiming Liu, Professor, Beijing Tiantan Hospital
Other Study IDs: HX-B-2022062
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic subdural hematoma; Dietary inflammatory index; Food frequency questionnaire; Modified frailty index
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Diet; Nervous System Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Chronic subdural hematoma group:
  * vein blood
  * stool
  * urine
  * hematoma fluid
  * dura mater
  * hematoma outer membrane
  Healthy control group:
  * vein blood
  * stool
  * urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group (CSDH group): CSDH patients recruited from neurosurgical department at 4 medical centres in China, which have apparent clinical symptoms and are confirmed by computed tomography or magnetic resonance imaging.
  Interventions: Other: Dietary and nutritional questionnaire; Other: Neurological function, cognitive function, and life quality assessment; Other: Peripheral blood test; Other: Metabonomic test; Other: Hematoma test
- Control group (Healthy group): non-CSDH, age- and gender-matched patients recruited from ophthalmology, otolaryngology, and physical examination department at 4 medical centres in China.
  Interventions: Other: Dietary and nutritional questionnaire; Other: Peripheral blood test; Other: Metabonomic test

INTERVENTIONS:
Other: Dietary and nutritional questionnaire — Nutrition assessment, nutrient intake, dietary inflammatory index, and frailty status will be examined using questionnaires.
Other: Neurological function, cognitive function, and life quality assessment — Neurological function, cognitive function, and life quality will be examined using Glasgow Coma Scale, Modified Rankin Scale, Markwalder Grade Scale, Mini-mental state examination, and EuroQol five dimensions questionnaire.
  Groups: Case group (CSDH group)
Other: Peripheral blood test — Collect peripheral blood samples from patients.
Other: Metabonomic test — Collect urine and stool samples from patients.
Other: Hematoma test — Collect hematoma fluid, dura mater, and hematoma outer membrane samples from patients.
  Groups: Case group (CSDH group)

SUMMARY:
A prospective, multicenter, case control trial is designed to compare difference in dietary and nutritional factors in patients with and without chronic subdural hematoma.

DETAILED DESCRIPTION:
Chronic subdural hematoma (CSDH) is one of the most common neurosurgical conditions, which is considered to be an inflammatory disease. Dietary factors can have an impact on the inflammatory mechanism in human body, which can increase a variety of inflammatory biomarkers in the blood. The risk of malnutrition in the elderly is generally high, and nutritional status can affect the risk of CSDH in the elderly. Little is known about the association of dietary factors with CSDH. The investigators speculate that dietary factors participate in and promote the occurrence and development of CSDH. This study will clarify whether there is a correlation between dietary factors and CSDH, which will reveal the pathogenesis and prevention of CSDH.

ELIGIBILITY:
Case group (CSDH group)

Inclusion Criteria:

* Patients (18 years to 90 years) presenting with clinical symptoms and neurological deficits of CSDH.
* CSDH verified on cranial computed tomography or magnetic resonance imaging.
* Written informed consent from patients or their next of kin according to the patient's cognitive status.

Control group (Healthy group)

Inclusion Criteria:

* non-CSDH patients (18 years to 90 years) with matched age and gender.
* Written informed consent from patients or their next of kin according to the patient's cognitive status.

Exclusion Criteria for both case and control group:

* Previous intracranial surgery for any neurological disorders but chronic subdural hematoma before.
* CSDH turned from acute subdural hematoma.
* Existing malignant tumors, poor medication condition or severe comorbidity.
* Difficulty in feeding requiring long-term enteral or parenteral nutrition support.
* Dietary and nutritional survey is estimated to be completed difficultly.
* Reproductive-age women without verified negative pregnancy testing.
* Participating in other research.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CSDH patients and non-CSDH, age- and gender-matched patients recruited from 4 medical centres in China.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Difference in dietary intakes | When subjects are enrolled
  Difference in dietary intakes assessed by Food Frequency Questionnaire, a common method for measuring dietary intake in large epidemiological studies.
Difference in Dietary Inflammatory Index score | When subjects are enrolled
  The Dietary Inflammatory Index (DII) score of the current nutritional status of patients with and without CSDH will be evaluated. The amounts of nutrients will be calculated using last 3-month nutrient analysis program. DII score will calculate from these foods. The z-score must first be calculated. To calculate the z-score, the standard global consumption amount is subtracted from the average consumption amount of the individual. The result obtained is divided by the standard deviation value. The z score found with this result is converted to the percentile score. The percentile value is multiplied by the full inflammatory effect score. DII is obtained as a result of summing the scores calculated for all nutrients. Found DII is an indicator of the inflammatory load of the individual's daily diet.
Difference in nutritional status | When subjects are enrolled
  Difference in nutritional status measured by Mini-Nutritional Assessment.
Difference in frailty status | When subjects are enrolled
  Difference in frailty status measured by Modified Frailty Index. Modified Frailty Index ranges from score 0 to 1, and frail status is defined as a score of ≥0.27.

SECONDARY OUTCOMES:
Difference in gut microbiota measured by 16S rRNA between case group and control group | When subjects are enrolled
  Fecal sample will be measured by 16S rRNA sequencing. The alpha and beta diversity of gut microbiota between the groups will be analyzed, including a series of statistical analysis indexes such as Chao, Shannon, Simpsonace, Simpson and Coverage, in order to reflect the microbial community diversity. Based on the results of species annotation, the community histogram, the community heatmap and the Wayne map will be used to analyze the species composition of the sample, in order to explore the relationship between the species and the sample, and analyze the key microflora in the sample. The PCA, PCoA and NMDS analysis will be used to assess the similarities and differences in species composition between groups. To further screen the species with significant differences, the LEfSe difference discriminant analysis will be used.
Difference in metabolomics of gut, urine, and serum between case group and control group | When subjects are enrolled
  Changes of metabolites in gut, urine, and serum will be measured by metabolomic mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Liu, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (4):
- China (4):
  - Huangshan City People's Hospital, Huangshan City, Anhui
  - First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Beijing Tiantan Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No